CLINICAL TRIAL: NCT00078754
Title: Fluoxetine and Divalproex: Treatment Correlates in IED
Brief Title: A Comparison of Fluoxetine and Divalproex for the Treatment of Intermittent Explosive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH066984 (NIH); R01MH066984 (NIH); DATR A5-ETMA
Record Dates: First submitted 2004-03-05; First posted 2004-03-08 (Estimated); Results first posted 2014-12-31 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Intermittent Explosive Disorder
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders | interventions — Fluoxetine; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Participants will to receive treatment with fluoxetine for 12 weeks
  Interventions: Drug: Fluoxetine
- B (Experimental): Participants will to receive treatment with divalproex for 12 weeks
  Interventions: Drug: Divalproex
- C (Placebo Comparator): Participants will to receive treatment with placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine — Fluoxetine capsules by mouth, up to 60 mg daily
  Arms: A
Drug: Divalproex — Divalproex ER capsules by mouth, up to 3000 mg daily
  Arms: B
Drug: Placebo — Placebo capsules by mouth, up to 8 capsules daily
  Arms: C

SUMMARY:
This study will compare the medications fluoxetine (Prozac®) and divalproex (Depakote®) for the treatment of aggressive behavior in individuals with Intermittent Explosive Disorder (IED).

DETAILED DESCRIPTION:
IED is a condition characterized by a failure to resist aggressive impulses. IED is a behavioral defined condition for which effective treatments have not been identified. Research suggests that serotonin (5-HT), a chemical that helps regulate mood and emotions, may play a role in the response to pharmacological IED treatments. This study will examine the relationship between 5-HT receptors and response to treatment with fluoxetine or divalproex. In addition, this study will examine people with IED and those without the condition to determine whether there are differences in their 5-HT receptor and transporter systems.

Participants in this study will be randomly assigned to receive either fluoxetine, divalproex, or placebo for 12 weeks. Scale ratings will be used to assess the aggression levels of participants. Biologic evaluations of the 5-HT system will be conducted throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Intermittent Explosive Disorder (IED)
* In good physical health
* Overt Aggression Scale-Modified (OAS-M) score of 15 or higher at screening
* Willing and able to comply with the study requirements

Exclusion Criteria:

* Life history of bipolar disorder, schizophrenia, organic mental syndrome, or mental retardation
* Current major depressive disorder, with a Hamilton Depression (HAM-D) Scale score higher than 18
* Current alcohol or drug abuse or dependence
* Active medical conditions that will interfere with the study
* Thymoleptic or neuroleptic treatments
* Presence of the following serious and active medical conditions: demyelinating or progressive degenerative disorders; central nervous system infection; progressive degenerative neurological disorder; ischemic heart disease; respiratory, renal, or liver disease; Type I diabetes; malignant neoplasm; hyper- or hypo-coagulopathy; Acquired Immune Deficiency Syndrome (AIDS); or seizure disorder. Participants with a history of more than two febrile seizures prior to 1 year of age are eligible.
* Chronic, ongoing treatment with the following classes of medications: antidepressants, neuroleptics, mood stabilizers, antianxiety agents, hypnotics, narcotics or synthetic narcotics, barbiturates, stimulants, anti-migraine agents, anti-epileptics, non-beta-blocking or Ca-channel blocking anti-arrhythmic agents prescribed to treat cardiac arrhythmia, anticoagulants, immunomodulators, anti-neoplastic agents, or HIV antiviral agents
* Ongoing psychotherapeutic treatment for the treatment of IED or anger that was started less than 3 months before study entry
* Hypersensitivity to fluoxetine or divalproex
* Pregnancy

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2003-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emil F. Coccaro, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A - Fluoxetine Drug: Participants will to receive treatment with fluoxetine for 12 weeks
  Fluoxetine: Fluoxetine capsules by mouth, up to 60 mg daily
- Group B - Divalproex Drug: Participants will to receive treatment with divalproex for 12 weeks
  Divalproex: Divalproex ER capsules by mouth, up to 3000 mg daily
- Group C - Placebo: Participants will to receive treatment with placebo for 12 weeks
  Placebo: Placebo capsules by mouth, up to 8 capsules daily
Period: Overall Study
Arm/Group | Group A - Fluoxetine Drug | Group B - Divalproex Drug | Group C - Placebo
Started | 29 | 30 | 31
Completed | 14 | 11 | 16
Not Completed | 15 | 19 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A - Fluoxetine Drug | Group B - Divalproex Drug | Group C - Placebo | Total
Number analyzed (Participants) | 29 | 30 | 31 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 30 | 31 | 90
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 16 | 40
  Male | 15 | 20 | 15 | 50
overt aggression scale-modified (OAS-M). [Mean (Standard Deviation); unit: units on a scale] — OAS-M is a validated instrument that measures aggression. Possible scores for aggression range from 0 (no aggression) to infinity (because the score is calculated by the number of times an aggressive behavior occurred, which theoretically has no possible maximum). Therefore the bigger number, the more aggression. OAS-M score was calculated for the past week before the visit.
  units on a scale | 36.75 (46.88) | 36.96 (26.42) | 66.08 (77.99) | 47.30 (56.68)

OUTCOME MEASURES:

1. Primary Outcome: Overt Aggression Scale-Modified for Outpatient Use (OAS-M)
Description: OAS-M is a validated instrument that measures aggression. Anti-aggressive effect of the drug/placebo was measured by the aggression score from OAS-M. Possible scores for aggression range from 0 (no aggression) to infinity (because the score is calculated by the number of times an aggressive behavior occurred, which theoretically has no possible maximum). Therefore the bigger number, the worse anti-aggression effect, thus the worse outcome. In each weekly visit, OAS-M score was calculated for the past week.
Time Frame: Measured at Week 12
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Fluoxetine Drug | Group B - Divalproex Drug | Group C - Placebo
Number analyzed (Participants) | 14 | 11 | 16
units on a scale | 7.86 (4.11) | 15.73 (10.15) | 8.88 (3.51)
Statistical Analysis 1: Comparison: Group A - Fluoxetine Drug vs Group B - Divalproex Drug vs Group C - Placebo; Test type: Superiority or Other; p = 0.622, ANCOVA

2. Secondary Outcome: OAS-M
Description: Overt Aggression Scale Modified for Outpatient Use. Minimum value = 0 Maximum value = Infinity. Higher scores means worse outcome.
Time Frame: Measured at Week 12
Population: OAS-M Scores in Placebo, Fluoxetine, Divalproex Arms as a function of LHA Score.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Fluoxetine: 20-60 mg po qd for up to 12 weeks.
- Divalproex: Up to 3000 mg po qd for up to 12 weeks.
- Placebo: Up to 8 capsules po qd for up to 12 weeks.
Arm/Group | Fluoxetine | Divalproex | Placebo
Number analyzed (Participants) | 29 | 30 | 31
score on a scale
  High Aggression Group: number analyzed (Participants) | 20 | 22 | 21
  High Aggression Group | 13.2 (5.0) | 13.7 (4.8) | 19.5 (5.1)
  Medium Aggression Group: number analyzed (Participants) | 9 | 8 | 10
  Medium Aggression Group | 25.1 (7.6) | 29.6 (8.0) | 26.9 (7.1)
Statistical Analysis 1: Comparison: Fluoxetine; The hypothesis was that subjects with LHA Scores = 18 or more would respond better to divalproex (than fluoxetine) while those with LHA scores = or < 17 would respond better to fluoxetine (than divalproex); Test type: Superiority; p = 0.029, ANCOVA — LHA score main effect; The LHA Score F[1,83] = 4.91, p = 0.029; Condition F[2,83] = 0.20, p = 0.815; Condition x LHA Score F[2,83] = 0.255, p = 0.799
Statistical Analysis 2: Comparison: Fluoxetine vs Divalproex; ANCOVA at endpoint with baseline OAS-M AGG score as covariate; Test type: Superiority; p = 0.80, ANCOVA; Baseline OAS-M Aggression score as covariate; Mean Difference (Final Values) = 19.0, Standard Error of Mean 2.7

ADVERSE EVENTS:
Arm/Group | Group A - Fluoxetine Drug | Group B - Divalproex Drug | Group C - Placebo
Serious Adverse Events (participants affected / at risk) | 1/29 | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 23/29 | 23/30 | 24/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A - Fluoxetine Drug (N=29) | Group B - Divalproex Drug (N=30) | Group C - Placebo (N=31)
hyponatremia/hypokalemia (Blood and lymphatic system disorders) | 1 | 0 | 0 — lab results showed hyponatremia/hypokalemia.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A - Fluoxetine Drug (N=29) | Group B - Divalproex Drug (N=30) | Group C - Placebo (N=31)
Headaches (Investigations) | 7 | 6 | 8
Trembling (Investigations) | 2 | 3 | 1
Faintness or dizziness (Investigations) | 2 | 3 | 4
Numbness or tingling in parts of your body (Investigations) | 5 | 4 | 3
Feeling tense or keyed up (Investigations) | 14 | 11 | 14
Nervousness or shakiness inside (Investigations) | 6 | 6 | 4
Soreness in your muscle, back, joints (Investigations) | 13 | 17 | 16
Spells of terror or panic (Investigations) | 2 | 3 | 2
Hot or cold spells (Investigations) | 3 | 6 | 4
Heart pounding or racing (Investigations) | 6 | 6 | 5
Pains in the heart or chest (Investigations) | 2 | 4 | 2
Trouble getting your breath (Investigations) | 1 | 6 | 6
Trouble remembering things (Investigations) | 9 | 6 | 7
Feeling that familiar things are strange or unreal (Investigations) | 2 | 4 | 0
Nausea or upset stomach (Investigations) | 5 | 9 | 9
Drowsiness (Investigations) | 8 | 12 | 10
Dry mouth (Investigations) | 5 | 9 | 4
Blurred vision (Investigations) | 2 | 2 | 2
Increased salivation (Investigations) | 1 | 4 | 2
Sweating (Investigations) | 6 | 9 | 4
Diarrhea (Investigations) | 2 | 5 | 5
Difficulty urinating (Investigations) | 1 | 1 | 1

LIMITATIONS AND CAVEATS:
Most participants did not have stable OAS-M Aggression scores from screening to randomization. Note that this was not a requirement for this study; only that OAS-Aggression scores were 15 or higher at screening.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No